CLINICAL TRIAL: NCT04756986
Title: Efficacy of Malic Acid Spray in Treatment of Xerostomia in Type II Diabetic Patients
Brief Title: Malic Acid in Treatment of Xerostomia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Malic acid in xerostomia
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia | interventions — malic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- malic acid group (Experimental): patients will receive a topical spray containing 1% malic acid
  Interventions: Drug: malic acid
- placebo group (No Intervention): patients will receive a topical placebo spray

INTERVENTIONS:
Drug: malic acid — 1% malic acid spray
  Other Names: hydroxybutanoic
  Arms: malic acid group

SUMMARY:
Background: xerostomia is a subjective sensation of dry mouth resulting from quantitative and /or qualitative changes of saliva. Patients receiving drugs like antihypertensives and antidepressants or patients receiving chemotherapy or radiotherapy for treatment of head and neck cancers may suffer from xerostomia. It also can be experienced in patients with systemic diseases like diabetes mellitus, systemic lupus erythematosus, sjogren's syndrome and rheumatoid arthritis. Malic acid spray with concentration of 1% has grabbed the attention over the last few years as an effective treatment for xerostomia.

Study objective: To evaluate the effect of 1% malic acid spray in treatment of xerostomia in type 2 diabetic patients.

DETAILED DESCRIPTION:
This randomized controlled clinical trial included 52 patients with type 2 diabetes mellitus suffering from xerostomia, divided equally into two groups. Group-I was managed by topical spray containing 1% malic. Group- II was managed by a placebo spray. Both groups received the treatment for 2 weeks. Dry mouth questionnaire scores (DMQ) and unstimulated salivary flow rate was collected before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus suffering from xerostomia.
* Patients aged between 35 and 50 years old.
* Glycated hemoglobin less than 7% (28) .
* Duration of diabetes mellitus not less than 4 years and not more than 8 years.

Exclusion Criteria:

* Patients receiving any drugs that cause hyposalivation like anti-hypertensive drugs.
* Patients with any systemic disease reported to produce hyposalivation (sjogren's syndrome, hepatitis c, rheumatoid arthritis and lupus erythematosus) (8).
* Patients receiving chemo-therapy and radio-therapy.
* Mouth breathers.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
The unstimulated salivary flow rate | 4 weeks
  The unstimulated salivary flow rate will be obtained by the spit method every 30s for 15 minutes. Saliva will be collected in graduated tubes. Measurements will be expressed as milliliter per minute. Participants will be asked to refrain from eating, drinking and brushing their teeth at least 2 hours before saliva collection
  - Hypo-salivation if the unstimulated salivary flow rate 0.1- 0.2 ml/min or less

SECONDARY OUTCOMES:
scoring of severity of xerostomia | 4 weeks
  Each individual's responses will be scored and summed to give a single score and the higher scores represent more severe symptoms using Xerostomia Inventory-Dutch version

CONTACTS AND LOCATIONS:
Overall Officials: Eglal M Mousa, PHD, Study Director — Alexandria University; Yasmin Y Gaweesh., PHD, Principal Investigator — Alexandria University; Noha K. Abo Aasy, PHD, Principal Investigator — Alexandria University; Shaimaa A. Muhamed, BDS, Principal Investigator — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The investigators are planning to share the methods and the results of this study with all the investigators
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication
Access Criteria: he sharing access can be through PubMed when the study is published or through direct contact through this email